CLINICAL TRIAL: NCT03348124
Title: Prevention of Unwanted Pregnancy and a Path to Informed Choice Among Young People With Intellectual Disability- a RCT, Intervention With Conversational Support and Real-Care-Baby Simulator
Brief Title: Prevention Among Young People With Intellectual Disability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Uppsala University (Other)
Collaborators: Uppsala-Örebro Regional Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Prevention ID
Record Dates: First submitted 2017-11-10; First posted 2017-11-20 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Intellectual Disability; Adolescent Development; Young Adult
Keywords: Intellectual disability; Parenthood; Reproduction; Intervention; Adolescents
MeSH Terms: conditions — Intellectual Disability | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Cluster randomized intervention study with waiting list control group.
Who Masked: Outcomes Assessor
Masking Description: The researchers are outcome assessors, independent from the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Educational lessons based on the conversational material Toolkit "Children - what does it involve?", will be delivered in the classroom at school and caring for the RCB simulator during three days and nights.
  Interventions: Behavioral: "Children - what does it involve?"
- Control (No Intervention): Education as usual.

INTERVENTIONS:
Behavioral: "Children - what does it involve?" — Thirteen educational lessons based on the conversational material Toolkit will be delivered in the classroom at school, two lessons per theme. The themes consists of: 1) a card game: "What i wish" 2) Time 3) Money 4) Skills 5) Relations 6) Housing. The material is prepared and same for all schools. This intervention will be given 1-2 lessons per week over a period of 8-14 weeks. During this period the students also care for the RCB simulator during three days and nights, but with a break for "day care" for the simulator which was between 7 am and 5 pm when the students were in school. All students will practice handling the simulator to be familiar with all types of needs: to rock, change diaper, feed and burp and were taught the skills of head support, techniques to avoid rough handling.
  Other Names: education as usual
  Arms: Intervention

SUMMARY:
This study aims to evaluate an intervention using the Toolkit "Children - what does it involve?" and the "Real-Care-Baby" (RCB) simulator among students with intellectual disability (ID), using a cluster randomized trial design with waiting-list control group.

DETAILED DESCRIPTION:
Background: There is limited knowledge about how young people with ID can be facilitated in their process of deciding about parenthood. A feasibility study showed that it is possible to evaluate an intervention using the chosen instruments among students with ID in order to provide them with further insights about parenthood. Methods: Randomization of eleven clusters/schools to intervention and eleven clusters to waiting-list control. Intervention includes thirteen educational lessons and a three-day and night caring-session with the RCB simulator. Intervention will be given 1-2 lessons/week during 8-14 weeks. Data will be collected with questionnaires and interviews before and after intervention. In control group: Before and after waiting-list time and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Students with mild or moderate ID with informed consent can be included
* Understand and respond to a questionnaire

Exclusion Criteria:

- Students with severe ID

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Infant Simulator Attitude Scale (ISA) | Change from baseline after 13 weeks
  The original ISA consists of 38 items of which most are statements with four response alternatives ranging from strongly agree to strongly disagree. It was translated to Swedish and to the cognitive level of students with intellectual disability. Statements were changed into questions and one response alternative "I do not know" was added. The items related to sexual activity and to contraception were omitted since it was not the focus of the intervention and also to ease the all over burden of lengthy questionnaires for the students.

SECONDARY OUTCOMES:
General Self-Efficacy Scale (S-GSE) | Change from baseline after 13 weeks
  The S-GSE contains 10 items and it has already been used in Sweden. The investigators adapted two of the items and added the response alternative "I do not know". The layout of the response alternatives was adapted to individuals with cognitive disability and the students were given the opportunity to use pictures or sign language for ease of understanding.
Data extracted from Real Care Baby simulator | Change from baseline after three days and nights
  Proper care, mishandle and performance - mean and range in percent

CONTACTS AND LOCATIONS:
Overall Officials: Berit Höglund, PhD, Principal Investigator — Uppsala University Sweden
Locations (1):
- Uppsala Special school, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No